CLINICAL TRIAL: NCT02998723
Title: Does an Early Booster Session Improve Performance and Retention of Skills in Basic Life Support Compared to a Later Booster? A Simulation Based Randomized Controlled Trial
Brief Title: Early or Late Booster for Basic Life Support?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20150174-01H
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Basic Life Support
Keywords: Basic Life Support; Education, Medical; Cardiopulmonary Resuscitation; Learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early Booster Teaching (Experimental): The early booster group will receive a booster teaching session at 3 weeks post-training followed by feedback.
  Interventions: Other: Early Booster Teaching
- Late booster Teaching (Active Comparator): The late booster group will receive a booster teaching session at 2 months post-training followed by feedback.
  Interventions: Other: Late Booster Teaching
- Control group (No Intervention): The control group will receive no booster at all.

INTERVENTIONS:
Other: Early Booster Teaching — The early booster group will receive a booster teaching session at 3 weeks post-training followed by feedback.
  Arms: Early Booster Teaching
Other: Late Booster Teaching — The late booster group will receive a booster teaching session at 2 months post-training followed by feedback
  Arms: Late booster Teaching

SUMMARY:
Attrition of skills after basic life support (BLS) training is common. Psychology studies have established that for basic memory recall tasks, spaced learning strategies improve retention. Spaced learning is often organized as a refresher or 'booster' course after initial training. This study aims to investigate if this principle holds true for BLS skills, which require rapid memory recall and efficient deployment of procedural skills while under time pressure.

DETAILED DESCRIPTION:
Novice laypeople who have not received BLS training in the 6 months leading up to the date of participation will be recruited from the University of Ottawa and the general public. Participants will be randomized into one of three groups: early booster, late booster, or no booster (control). Currently, no booster is the educational standard. The early booster group will receive a booster at 3 weeks, the late booster at 2 months, and no booster for the control. All participants will undergo BLS training, an immediate post-test, and a retention post-test at 4 months. Post-tests involve a simulated cardiac arrest scenario. Raters will be blinded to the group allocation and simulation test order.

ELIGIBILITY:
Inclusion Criteria:

* Laypeople who have not received any BLS training or practice in the 6 months leading up to the date of their participation will be recruited.

Exclusion Criteria:

* Under 18 years old;
* Non layperson and Basic Life Training in less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Basic Life Support performance, as measured by the standardized Heart and Stroke Heartsaver checklist | 4 months
  BLS performance, as measured by the standardized Heart and Stroke Heartsaver checklist

SECONDARY OUTCOMES:
Time to start chest compression; | 4 months
  Time from entering the scene to initiation of compression (in seconds)
Accuracy of compression depth | 4 months
  Percentage of compressions that are deep enough
Compression ratio | 4 months
  The percentage of time during the scenario that compressions are done
Hand position | 4 months
  The percentage of time the hand position is correct
Tidal volume | 4 months
  Mean tidal volume (ml)
Ventilation success rate | 4 months
  The percentage of time ventilations are done with adequate volume 400-700mls
Time to defibrillation using AED. | 4 months
  Time from start to defibrillation using AED (in seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boet S, Waldolf R, Bould C, Lam S, Burns JK, Moffett S, McBride G, Ramsay T, Bould MD. Early or late booster for basic life support skill for laypeople: a simulation-based randomized controlled trial. CJEM. 2022 Jun;24(4):408-418. doi: 10.1007/s43678-022-00291-3. Epub 2022 Apr 19. PMID 35438450